CLINICAL TRIAL: NCT03102151
Title: Reducing the Duration of Untreated Psychosis Through Community Education
Brief Title: Reducing the Duration of Untreated Psychosis
Acronym: ReduceDUP
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven R. Lopez, Professor, University of Southern California
Other Study IDs: USCLaCLAVE; 1R01MH103830 (NIH)
Record Dates: First submitted 2016-08-01; First posted 2017-04-05 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Community Campaign La CLAVE — A community campaign to teach community residents and professional networks the signs and symptoms of psychosis using social media, community talks, and advertising.

SUMMARY:
The study examines the possible effect of a community campaign to decrease the duration of untreated psychosis in persons with their first episode of a psychotic disorder.

DETAILED DESCRIPTION:
The study examines whether a community campaign can reduce over time the duration of untreated psychosis (DUP) among persons with first episode psychosis (FEP). The DUP of mental health patients with FEP who sought services at a public outpatient or an inpatient facility was assessed for a 15 month period prior to the campaign launch. This serves as the baseline or historical control. The DUP will continue to be assessed for another 3 years. The hypothesis being tested is that there will be a significant decrease in DUP between baseline, one-year, two-year and three-year follow-ups. This study is being carried out with Latinos in Los Angeles County because as a group, particularly among Spanish-speaking immigrants, Latinos are at high risk for prolonged DUP.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual-4 criteria for a psychotic disorder
* of Latino origin

Exclusion Criteria:

* has a neurological disorder or suffers from brain trauma

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Living in the catchment area of San Fernando Mental Health Outpatient clinic, a clinic with the Los Angeles County Department of Mental Health
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Latency to Treatment (LTT) a novel interview based assessment tool to measure the Duration of Untreated Psychosis | At the time of recruitment into the study
  The time from the onset of psychosis to the time the subject receives appropriate mental health treatment. The metric is number of weeks that the person went without treatment from illness onset. The number of weeks is the variable of interest that will be aggregated.

SECONDARY OUTCOMES:
Psychosis literacy, a questionnaire based inquiry for which the respondents answer either open-ended questions (e.g., What is serious mental Illness?) or "Yes-no" questions ("e.g., Can you recognize a serious mental illness in others?) | At the time of recruitment in to study
  The responses to the interview are either written down or audio-recorded. Raters then listen or read the responses and code them. The responses are aggregated as frequencies (e.g., the number of symptoms identified) or as percentages (e.g., the proportion of respondents who reported that they can recognize a serious mental illness in others).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lopez, PhD, Principal Investigator — University of Southern California
Locations (1):
- San Fernando Mental Health Center, Granada Hills, California, United States

IPD SHARING:
Plan to Share IPD: No